CLINICAL TRIAL: NCT00921973
Title: A Multicenter, Double-Blinded, Randomized, Placebo Controlled Study to Investigate the Safety and Immunogenicity of VAX102 When Given in the Same Arm With the Standard Influenza Vaccine in Healthy Adults
Brief Title: Safety of VAX102 Vaccine Given With Seasonal Flu Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAX102-07
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: influenza; universal influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — VAX102 vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAX102 (Active Comparator): Simultaneous administration of VAX102 1 ug i.m. plus TIV
  Interventions: Biological: VAX102
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VAX102 — All subjects receive TIV, one half of the subjects are randomized to receive VAX102 1 ug and one half are randomized to receive placebo
  Other Names: Universal influenza vaccine
  Arms: VAX102
Biological: Placebo — All subjects receive TIV, one half of the subjects are randomized to receive VAX102 1 ug and one half are randomized to receive placebo
  Arms: Placebo

SUMMARY:
The study will assess the safety, reactogenicity, and tolerability of VAX102 when given with Trivalent Inactivated Influenza Vaccine (TIV) delivered in the same arm as two separate IM injections in healthy adults 18 to 49 years. The investigators will measure the immunogenicity of the VAX102 when given with TIV and the antibody response to TIV when given with VAX102 compared to TIV alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 49 years inclusive
* Give written informed consent to participate in the study and adherence to all protocol requirements.
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations
* Females willing to practice birth control during the study.
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of vaccination.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
* Did not receive influenza vaccination (TIV) during the 2008-2009 influenza season.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness (institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months) as determined by medical history and/or physical exam.
* History of cancer.
* History of impaired immunoresponsiveness, including diabetes.
* Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs or any components of the study vaccines.
* Received influenza vaccination during the 2008-2009 season
* History of systemic hypersensitivity reactions to egg proteins, or any other component of FLUVIRIN®, or life-threatening reactions to previous influenza vaccinations.
* Has known history of Guillain-Barré Syndrome
* Presently receiving or history of receiving any medications or treatments that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months. Inhaled and topical corticosteroids will be allowed.
* Participated in a clinical trial or received or planned administration of an investigational compound within 30 days before receiving study vaccine and/or during the study through the Day 28 evaluation.
* Was vaccinated with a registered vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to receiving the study vaccine.
* History of anaphylactic type reaction to injected vaccines.
* History of drug or chemical abuse in the year before the study.
* Use of new prescription medications started within 7 days before study entry.
* Receipt of any blood products, including immunoglobulin, within 6 months before administration of study vaccine or anticipated receipt during the study period.
* Donation of blood or blood products within 8 weeks before study entry or at any time during the study.
* Has clinical signs of active infection and/or oral temperature of ≥ 38 (100.4 ºF). Study entry may be deferred for such individuals at the discretion of the investigator.
* Has evidence or history of (within the previous 12 months) drug or alcohol abuse.
* Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Immune response | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David N Taylor, MD, Study Director — VaxInnate Corporation
Locations (2):
- United States (2):
  - Johnson County Clin Trials, Lenexa, Kansas
  - Vanderbilt Clinical Trials Center, Nashville, Tennessee

REFERENCES:
- [Derived] Talbot HK, Rock MT, Johnson C, Tussey L, Kavita U, Shanker A, Shaw AR, Taylor DN. Immunopotentiation of trivalent influenza vaccine when given with VAX102, a recombinant influenza M2e vaccine fused to the TLR5 ligand flagellin. PLoS One. 2010 Dec 28;5(12):e14442. doi: 10.1371/journal.pone.0014442. PMID 21203437